CLINICAL TRIAL: NCT00909584
Title: Phase 2 Randomized Study of Ezatiostat Hydrochloride (Telintra™, TLK199 Tablets) for Treatment of Severe Chronic Neutropenia
Brief Title: Study of Ezatiostat (Telintra Tablets) for Treatment of Severe Chronic Neutropenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study TLK199.2103 was terminated for business reasons.
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.2103
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Severe Chronic Neutropenia
Keywords: Hematology; Neutropenia; SCN; Severe Chronic Neutropenia; Idiopathic; Telintra; ezatiostat hydrochloride; ezatiostat; TLK199; Glutathione; Glutathione analog; Glutathione Transferase; Glutathione Transferase inhibitor; Glutathione Transferase P1-1 inhibitor; GSTp1-1 inhibitor; Apoptosis; Differentiation; Enzyme inhibitor
MeSH Terms: conditions — Neutropenia, severe chronic; Neutropenia | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4-Week dose equilibration period with Telintra followed by 4 month treatment period
  Interventions: Drug: Ezatiostat Hydrochloride
- 2 (No Intervention): 4 Month observation period with standard of care treatment and option to crossover to Telintra treatment for 4 week dose equilibration followed by 4 week treatment period

INTERVENTIONS:
Drug: Ezatiostat Hydrochloride — Starting Dose 2000 mg orally per day in two divided doses with dose to increase or decrease to achieve target median ANC (Range 1,500-10,000 cells/uL)
  Other Names: Telintra tablets; TLK199 Tablets
  Arms: 1

SUMMARY:
This is a multicenter Phase 2 randomized parallel-group study to determine the effect of Telintra treatment on severe chronic neutropenia. Patients will be randomized to Telintra or enter an observation period with an option to crossover to Telintra treatment in a 1:1 allocation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Idiopathic Severe Chronic Neutropenia
* ECOG performance status of 0-2
* Adequate liver and renal function
* Adequate Red Blood Cell and Platelet counts

Exclusion Criteria:

* Prior treatment of SCN
* Non-Idiopathic types of SCN, ie. cyclic, congenital
* History of chromosomal abnormalities, myelodysplasia, hematologic malignancy, aplastic anemia, systemic lupus erythematosus, rheumatoid arthritis (Felty's syndrome), or other collagen diseases, and drug-induced neutropenia, autoimmune neutropenia
* Use of granulocyte colony stimulating factors (G-CSF), glucocorticoids, gamma globulin, lithium or investigational drug(s) within one month of enrollment
* History of bone marrow transplantation or stem cell support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Objective absolute neutrophil count (ANC) response rate | 18 Months

SECONDARY OUTCOMES:
Incidence of infections, oropharyngeal ulcers and antibiotic use | 18 Months
Incidence and duration of hospitalizations | 18 Months
FACT-N quality of life assessment | 18 Months
Safety assessments | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gail Brown, MD, Study Director — Telik
Locations (4):
- United States (4):
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington